CLINICAL TRIAL: NCT05558618
Title: Analysis of Personality Characteristics and Psychological Capital Factors on the Leadership of Pediatric Clinical Nurses
Status: Completed | Type: Observational
Sponsor: Hunan Children's Hospital (Other Government)
Responsible Party: Principal Investigator, xie jianhui, Director, Hunan Children's Hospital
Other Study IDs: HCHospital 001
Record Dates: First submitted 2022-09-21; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Pediatric Nursing; Leadership

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Survey Methods In this study, a questionnaire on nursing leadership and influencing factors was distributed online through Wenjuanxing, an online questionnaire platform. The nursing department and the head nurse of the department where the questionnaire was to be distributed were first contacted and they agreed, and the researcher joined each department's nurses' WeChat group, distributed the questionnaire QR code, and explained the inclusion and exclusion criteria and the method of completing the questionnaire, emphasizing that the questionnaire was filled in anonymously. Nurses in each department were given 24 hours to participate in the response (the response time was around 30 minutes).

Quality Control The selected nursing leadership questionnaire, EPQ-RSC scale and psychological capital questionnaire all had good reliability and validity; the inclusion and exclusion criteria and the method of completing the questionnaire were explained by the researcher to the participated nurses; questionnaires that were not filled out completely or filled out with obvious regularity, and those with L scores greater than 60 on the personality trait scale were considered invalid and were excluded; the data were checked by two people after collection.

Statistical methods SPSS 22.0 was used for statistical analysis. Continuous-type data were described using the mean ± standard deviation ( ), and single-sample t-test was used for those satisfying normal distribution. Count data were described using frequency and composition ratios. Dichotomous logistic regression was used to analyze the factors influencing the leadership of pediatric clinical nurses; P<0.05 was considered a statistically significant difference when not specifically stated.

ELIGIBILITY:
Inclusion Criteria:

* registered nurses working in clinical practice;
* those who voluntarily participated in this study.

Exclusion Criteria:

* those who did not work in the hospital during the survey period or who had not been on duty for ≥ 3 months in the past 1 year.

Ages: 23 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: nurses from 4 medical institutions in Hunan Province
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Gender of the subjects | 24 hour
  It contains 122 female subjects
Age of the subjects | 24 hour
  All 122 subjects were aged 23 to 55 (36.16 ± 6.75) years
Title of the subjects | 24 hour
  There were 69 nurses (56.6%) in secondary hospitals and 53 (43.4%) in tertiary hospitals
Have attended leadership courses or training | 24 hour
  68 nurses (55.7%) had attended leadership courses or training and 54 nurses (44.3%) had not attended leadership courses or training
Mean scores of dimensions and items of pediatric clinical nurse leadership | 24 hour
  The total score of leadership of pediatric clinical nurses was 181.48±26.43, with a mean score of 3.95±0.57, and the items in each dimension were problem solving ability, professional nursing ability, planning and organizing ability, communication ability, critical thinking ability, interpersonal ability, and self-care ability in order of mean score
Mean scores of the dimensions and items of personality traits of pediatric clinical nurses | 24 hour
  The items of personality traits of pediatric clinical nurses were psychoticism, neuroticism of the Pediatric Clinical Nurses Personality Trait Scale, extraversion and Lie. The average score of each item is 1.60±1.23, 7.55±2.95, 5.43±3.55, 6.79±1.96.
Mean scores of the dimensions and items of psychological capital of pediatric clinical nurses | 24 hour
  The total score of psychological capital of pediatric clinical nurses was 93.07±13.38, with a mean score of 4.55±0.67, and the items in each dimension were optimism, self-efficacy, resilience and hope.

CONTACTS AND LOCATIONS:
Locations (1):
- Jian-Hui Xie, Changsha, Hunan, China